CLINICAL TRIAL: NCT07002905
Title: A Phase IIa, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy, Safety, and Tolerability of ASC30 Tablets and ASC30 Tablets A1 in Participants With Obesity or Overweight With Weight-Related Comorbidities
Brief Title: A Study to Evaluate the Efficacy, Safety, and Tolerability in Participants With Obesity or Overweight With Weight-Related Comorbidities
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ascletis Pharma (China) Co., Limited (Industry)
Responsible Party: Sponsor
Organization: Ascletis Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ASC30-202
Record Dates: First submitted 2025-05-15; First posted 2025-06-04 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Chronic Weight Management

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Cohort 1 (Experimental): Participants will receive ASC30 tablets/ASC30 tablets A1 or Placebo administered orally once daily.
  Interventions: Drug: ASC30 tablets or ASC30 tablets A1 or placebo
- Cohort 2 (Experimental): Participants will receive ASC30 tablets/ASC30 tablets A1 or Placebo administered orally once daily.
  Interventions: Drug: ASC30 tablets or ASC30 tablets A1 or placebo
- Cohort 3 (Experimental): Participants will receive ASC30 tablets/ASC30 tablets A1 or Placebo administered orally once daily.
  Interventions: Drug: ASC30 tablets or ASC30 tablets A1 or placebo
- Cohort 4 (Experimental): Participants will receive ASC30 tablets/ASC30 tablets A1 or Placebo administered orally once daily.
  Interventions: Drug: ASC30 tablets or ASC30 tablets A1 or placebo
- Cohort 5 (Experimental): Participants will receive ASC30 tablets/ASC30 tablets A1 or Placebo administered orally once daily.
  Interventions: Drug: ASC30 tablets or ASC30 tablets A1 or placebo
- Cohort 6 (Experimental): Participants will receive ASC30 tablets/ASC30 tablets A1 or Placebo administered orally once daily.
  Interventions: Drug: ASC30 tablets or ASC30 tablets A1 or placebo
- Cohort 7 (Experimental): Participants will receive ASC30 tablets/ASC30 tablets A1 or Placebo administered orally once daily.
  Interventions: Drug: ASC30 tablets or ASC30 tablets A1 or placebo

INTERVENTIONS:
Drug: ASC30 tablets or ASC30 tablets A1 or placebo — Drug: ASC30 tablets or ASC30 tablets A1 administered orally daily Drug: Placebo administered orally daily

SUMMARY:
This randomized, double-blind, placebo-controlled phase IIa study is designed to evaluate the efficacy, safety, and tolerability of ASC30 Tablets and ASC30 Tablets A1.

ELIGIBILITY:
Inclusion Criteria:

* Have provided informed consent before initiation of any study-specific procedures.
* Male or female participants, non-smokers, between 18 and 75 years of age (both inclusive).
* No clinically significant findings from medical history, physical examination, 12-lead ECG, vital signs measurements, and other screening procedures.

Exclusion Criteria:

* Have evidence of any clinically significant active or chronic disease.
* Have any prior diagnosis of diabetes mellitus (T1DM or T2DM), or rare forms of diabetes mellitus.
* Have an autoimmune disease, is immunosuppressed or is in any way immunocompromised.
* Have a history of acute or chronic pancreatitis.
* Participants with a known clinically significant gastric emptying abnormality.
* Have a history of an active or untreated malignancy or are in remission from a clinically significant malignancy.
* Have a history of any other condition (such as known drug or alcohol abuse, diagnosed eating disorder, or other psychiatric disorder) that, in the opinion of the Investigator, may preclude the participant from following and completing the protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2025-07-03 (Actual); Primary Completion 2025-12-08 (Actual); Study Completion 2025-12-08 (Actual)

PRIMARY OUTCOMES:
Percent change in body weight from Baseline up to Week 13 | Baseline and Week 13

SECONDARY OUTCOMES:
Change in body weight (absolute) from Baseline up to Week 13 | Baseline and Week 13
Change in waist circumference from Baseline up to Week 13 | Baseline and Week 13
Change in body mass index from Baseline to Week 13 | Baseline and Week 13
Treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) | Baseline and Week 13

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Ascletis Clinical Site, Rogers, Arkansas
  - Ascletis Clinical Site, Fort Myers, Florida
  - Ascletis Clinical Site, Miami, Florida
  - Ascletis Clinical Site, Columbus, Ohio
  - Ascletis Clinical Site, Bellaire, Texas
  - Ascletis Clinical Site, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No